CLINICAL TRIAL: NCT04517578
Title: European Neuromuscular Monitoring Survey
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: EUNeuroMuscMonitoringSurvey
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-07

CONDITIONS: Availability of the Different Types of Anesthesia Neuromuscular Monitoring Devices Throughout European Hospitals; Health Care Utilization; Medical Device Availability; Medical Staff Availability
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Participants will be asked to fill in an online survey that will be anonimized.

SUMMARY:
This survey aims to better define the availability of the different types of anesthesia neuromuscular monitoring devices throughout European hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Active Anesthesiology department heads of European Anesthesiology departments.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: anaesthesia departments within the European health system.
Sampling Method: Probability Sample
Enrollment: 692 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Questionnaire about medical equipment and staff availability | 1 year
  Questionnaire about all medical equipment and staff that is available site per site and what is mainly used.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Publication in a journal.